CLINICAL TRIAL: NCT02444130
Title: Presbyopia Compensation: Looking for Electrophysiological Predictors
Status: Completed | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-A01677-38
Record Dates: First submitted 2015-02-18; First posted 2015-05-14 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Presbyopia
Keywords: multifocality; monovision
MeSH Terms: conditions — Presbyopia | interventions — Contact Lenses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: contact lenses — Presbyopia was compensated with contact lenses by monovision and multifocality.

SUMMARY:
The main purpose of this study was to identify electrophysiological predictive markers of post-correction visual comfort for presbyopic patients.

DETAILED DESCRIPTION:
For each participant, presbyopia was compensated with contact lenses by monovision during three weeks and multifocality (three weeks again). A break of two weeks without any presbyopia compensation came in between the two phases of the test that were randomized.

All subjects were tested three times: before any compensation, after three weeks with monovsion and after three weeks with multifocality.

Each testing session was strictly the same including visual examinations and VEPs (visual evoked potentials).

ELIGIBILITY:
Inclusion Criteria:

* normal acuity

Exclusion Criteria:

* stereoacuity disorder
* neurological disorders

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with presbyopia
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity at baseline | baseline
  near and distance visual acuity (Monoyer and Parinaud scales)

SECONDARY OUTCOMES:
electrophysiological recordings at baseline | baseline
  monocular and binocular pattern Visual Evoked Potentials in response to a checkerboard pattern N75 and P100 components : amplitude, latency and topography
electrophysiological recordings change with monovision | after 3 weeks with monovision contact lenses
  monocular and binocular pattern Visual Evoked Potentials in response to a checkerboard pattern N75 and P100 components : amplitude, latency and topography
electrophysiological recordings with multifocality | after 3 weeks with multifocality contact lenses
  monocular and binocular pattern Visual Evoked Potentials in response to a checkerboard pattern N75 and P100 components : amplitude, latency and topography
quantitative measurement of stereopsis at baseline | baseline
  TNO plates
quantitative measurement of stereopsis with monovision | after 3 weeks with monovision contact lenses
  TNO plates
quantitative measurement of stereopsis with multifocality | after 3 weeks with multifocality contact lenses
  TNO plates
Visual acuity change with monovision | after 3 weeks with monovision contact lenses
  near and distance visual acuity (Monoyer and Parinaud scales)
Visual acuity change with multifocality | after 3 weeks with multifocality contact lenses
  near and distance visual acuity (Monoyer and Parinaud scales)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Jean Pisella, MD, PhD, Principal Investigator — University Hospital, Tours
Locations (1):
- University hospital Tours, Tours, France

REFERENCES:
- [Derived] Imbeau L, Majzoub S, Thillay A, Bonnet-Brilhault F, Pisella PJ, Batty M. Presbyopia compensation: looking for cortical predictors. Br J Ophthalmol. 2017 Feb;101(2):223-226. doi: 10.1136/bjophthalmol-2015-307581. Epub 2016 Apr 22. PMID 27107029